CLINICAL TRIAL: NCT02131285
Title: Stabilometric Assessment of Context Dependent Balance Recovery in Persons With Multiple Sclerosis: a Randomized Controlled Study
Brief Title: Stabilometric Assessment of Balance Recovery in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDG_Falls_01
Record Dates: First submitted 2014-04-24; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation,; Balance,; Sensory strategies,; Multiple Sclerosis,; Postural control
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Sensory training (Experimental): Experimental group received balance rehabilitation aimed at improving motor strategies and sensory strategies. Subjects in this group were treated to improve recovery of sensory impairment and were given exercises in the impaired sensory conditions, inhibiting the reliable sensory systems and forcing the Central Nervous System to use the impaired ones.
  Interventions: Other: Sensory training
- No sensory strategy (No Intervention): Control group received usual care rehabilitation which did not include training of sensory strategies.

INTERVENTIONS:
Other: Sensory training
  Arms: Sensory training

SUMMARY:
Background: Balance control relies on accurate perception of visual, somatosensory and vestibular cues. Sensory flow is impaired in Multiple Sclerosis (MS) and little is known about the ability of the sensory systems to adapt after neurological lesions reducing sensory impairment. The aims of the present study were to verify whether:

1. Balance rehabilitation administered in a challenging sensory conditions would improve stability in upright posture
2. the improvement in a treated sensory condition would transfer to a non treated sensory condition.

Methods: Fifty three persons with Multiple Sclerosis, median (min-max) Expanded Disability Status Scale score of 5 (2.5-6.5), participated in a Randomized Controlled Trial and were randomly assigned to two groups. The Experimental group received balance rehabilitation aimed at improving motor and sensory strategies. The Control group received rehabilitation treatment which did not include training of sensory strategies. Persons with Multiple Sclerosis were blindly assessed by means of a stabilometric platform with eyes open, eyes closed and dome, on both firm surface and foam. Anterior-posterior and medio-lateral sway, velocity of sway and the length of Center of Pressure (CoP) trajectory were calculated in the six sensory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or laboratory definite relapsing-remitting, primary or secondary progressive MS

Exclusion Criteria:

* Inability to stand independently in upright position for 30 seconds
* Inability to walk for 6 m even with an assistive device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline at three weeks (end of treatment) for the following variables: Length [mm]; Velocity[mm/s]; Sway[mm] | Baseline, 3 weeks (end of treatment)
  Multivariate assessment. Length [mm]: length of CoP trajectory computed as sum of CoP displacement on the platform surface for each frame; Velocity: velocity of oscillations along anterior-posterior (VelAP) and medio-lateral (VelML) axes. These are computed as the first time derivative of CoP AP and ML displacement.
  Sway: standard deviation of CoP time series along anterior-posterior (SwayAP) and medio-lateral (SwayML) axes;

SECONDARY OUTCOMES:
Number of falls | baseline, 3 weeks (end of treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Gnocchi ONLUS, Milan, Italy

REFERENCES:
- [Background] Cattaneo D, Jonsdottir J, Zocchi M, Regola A. Effects of balance exercises on people with multiple sclerosis: a pilot study. Clin Rehabil. 2007 Sep;21(9):771-81. doi: 10.1177/0269215507077602. PMID 17875557
- [Derived] Cattaneo D, Jonsdottir J, Regola A, Carabalona R. Stabilometric assessment of context dependent balance recovery in persons with multiple sclerosis: a randomized controlled study. J Neuroeng Rehabil. 2014 Jun 10;11:100. doi: 10.1186/1743-0003-11-100. PMID 24912561